CLINICAL TRIAL: NCT05124002
Title: Recombinant Human Adenovirus Type 5 Combined With Hepatic Artery Infusion Chemotherapy of FOLFOX in Patients With Intrahepatic Mass-forming Cholangiocarcinoma: a Single-site, Single-arm, Prospective Study
Brief Title: Recombinant Human Adenovirus Type 5 Plus HAIC of FOLFOX for Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21325-2-02
Record Dates: First submitted 2021-10-31; First posted 2021-11-17 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-08

CONDITIONS: Cholangiocarcinoma, Intrahepatic
Keywords: oncolytic virus; intrahepatic mass-forming cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Folfox protocol

STUDY DESIGN:
Intervention Model Description: HAIC (FOLFOX) + H101
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H101+HAIC (Experimental): Recombinant Human Adenovirus Type 5 (H101): intratumorally injected 3 days before HAIC. 1 vial (5.0 × 10^11 vp) if the maximum diameters of lesion ≤ 5 cm, 2 vials (1.0 × 10^12 vp) if the maximum diameters of lesion ≤ 10 cm, 3 vials (1.5 × 10^12 vp) if the maximum diameters of lesion is > 10 cm.
  HAIC (FOLFOX): Oxaliplatin 50 mg + 5-FU 1.5 g + leucovorin calcium
  Interventions: Drug: Recombinant Human Adenovirus Type 5; Drug: HAIC of FOLFOX

INTERVENTIONS:
Drug: Recombinant Human Adenovirus Type 5 — H101 will be intratumorally injected 3 days before HAIC. Dosage of H101: 1 vial (5.0 × 10^11 vp) if the maximum diameters of lesion ≤ 5 cm, 2 vials (1.0 × 10^12 vp) if the maximum diameters of lesion ≤ 10 cm, 3 vials (1.5 × 10^12 vp) if the maximum diameters of lesion is > 10 cm.
  Other Names: H101
Drug: HAIC of FOLFOX — Oxaliplatin 50 mg + 5-FU 1.5 g + leucovorin calcium. The infusion will be continued for 2-3 days according to patients' tolerance and tumor conditions. The standard treatment for HAIC consists of 4-6 cycles, with the second cycle being 3 weeks after the end of the first HAIC cycle and the subsequent cycles being 4 weeks after the end of the previous HAIC.
  Other Names: FOLFOX

SUMMARY:
Oncolytic viruses can selectively replicate in and destroy tumor cells. Recent studies indicate that recombinant human adenovirus type 5 (H101), which is the first approved oncolytic virus drug in the world, shows anti-tumor effects on liver cancer. This study aims to further verify the effect and safety of recombinant human adenovirus type 5 combined with HAIC in the treatment of intrahepatic mass-forming cholangiocarcinoma.

DETAILED DESCRIPTION:
This is a perspective, single-arm trial. According to previous studies, the PFS of HAIC for unresectable intrahepatic cholangiocarcinoma is approximately 8 - 10 months, and one year progression free rate is about 40%. We assumed that the study could detect 20% absolute difference and 1 year PFS rate could achieve 60% PFS by (FOLFOX + H101) over conventional HAIC (FOLFOX). Simon's two-stage design is used to estimate the sample size, with α value of 0.05 and power of 0.9. A total sample size of 66 participants are required.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, male or female
* Histologically or cytologically confirmed intrahepatic mass-forming cholangiocarcinoma (IMCC) with unresectable lesion(s) or patients who refuse surgery
* At least one measurable lesion according RECIST v1.1 criteria [spiral CT/MRI scan ≥ 10 mm (CT scan slice thickness no greater than 5 mm)]
* Life expectancy ≥ 3 months
* The function of vital organs meets the following requirements: absolute neutrophil count (ANC) ≥ 3.5 × 10^9/L; platelets ≥ 125 × 10^9/L; hemoglobin ≥ 8 g/dL; Serum albumin ≥ 2.8 g/dL; bilirubin ≤ 3 ULN, ALT/AST ≤ 2.5 ULN; ALT/AST in the presence of liver metastases ≤ 5 ULN; creatinine ≤ 1.5 ULN; euthyroid; LVEF > 50%
* The date of the first dose of study drug is ≥ 21 days from the date of previous anti-tumor treatment, and has recovered from adverse reactions to prior anti-tumor therapy to baseline or lower than grade 1 (according to CTCAE Version 5.0)(except alopecia)
* Female patients of childbearing potential (including early menopause, menopause < 2 years, and non-surgical sterilization), male patients and their partners must agree to use effective contraceptive measures during the study
* Patients or their legal representatives can understand and offer informed consent, being willing to take part in the follow-up with good compliance

Exclusion Criteria:

* Pregnant or lactating women, men or women who are reluctant to take effective contraceptive measures
* Previous treatment with oncolytic viruses (such as T-VEC)
* Abnormal coagulation function, or having a bleeding tendency, or receiving thrombolytic or anticoagulant therapy
* Patients with poor glycemic control
* Known central nervous system tumors, including metastatic brain tumors
* Accompanied by any unstable systemic diseases, including but not limited to severe infection, resistant hypertension, unstable angina, stroke or myocardial infarction within 6 months, congestive heart failure, and serious cardiac arrhythmia requiring medication, renal or metabolic disease requiring medication
* Known hypersensitivity to the study drug or oxaliplatin, leucovorin calcium, fluorouracil
* History of immunodeficiency or autoimmune disease, or receiving long-term systemic steroid therapy within 7 days before enrollment, or any form of immunosuppressive therapy
* Other conditions that are not suitable for participating in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 1 month
  The median amount of time from registration until disease progression or death, whichever occurs first. Disease progression was assessed via RECIST 1.1 criteria.

SECONDARY OUTCOMES:
1 year survival rate | 1 year
  The percentage of participants who are alive one year after the start of the treatment.
Objective response rate (ORR) | up to 1month
  The percentage of participants who have achieved either a complete or partial response, as assessed by Response Criteria in Solid Tumors (RECIST 1.1).
Disease control rate (DCR) | up to 1 month
  The percentage of participants who have achieved complete response, partial response and stable disease, as assessed by Response Criteria in Solid Tumors (RECIST 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: ZHANG YUEWEI, MD, Principal Investigator — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China